CLINICAL TRIAL: NCT05546775
Title: Immunological Profile and Clinical Characteristics of Children Diagnosed With Chronic Granulomatous Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jehan Mostafa Abd Alhameed, Immunological profile and Clinical characteristics of children diagnosed with chronic granulomatous disease, Assiut University
Other Study IDs: Immunological profile and CGD
Record Dates: First submitted 2022-08-30; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: CGD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DHR — To describe the clinical characteristics and pattern of presentation of patients diagnosed as CGD in Assiut, and to find the most common presenting symptoms.
  * To mention the immunological profile of patients diagnosed with CGD (Immunogloulins level - B, T, natural killer cells enumeration with flow cytometry- DHR123)
  * To assess the growth parameters in patients with CGD.

SUMMARY:
Immunological profile and Clinical characteristics of children diagnosed with chronic granulomatous disease

DETAILED DESCRIPTION:
CGD "chronic granulomatous disease is a rare genetically determined disorder aﬀecting the immune system characterized by recurrent and persistent bacterial and fungal infections due to the inability of the body's phagocytic cells (neutrophil and monocytes) to kill certain phagocytosed microorganisms.). CGD is caused by mutations in one of the ﬁve genes coding for NADPH(nicotinamide adenine dinucleotide phosphate ) oxidase subunits. Approximately 70% of cases are caused by mutations in the CYBB gene leading to X-linked CGD, which often causes a severe form of the disease. More than 700 pathogenic mutations in the CYBB gene encoding the gp91-phox protein have been documented. Other biallelic mutations in CYBA, NCF1, NCF2, and NCF4 cause autosomal recessive CGD. In addition, a novel ER-resident transmembrane protein called Eros (essential for reactive oxygen species) that is essential for the regulation of NADPH oxidase and controls the phagocyte respiratory burst was described. A homozygous CYBC1/EROS mutation was associated with the development of CGD Symptoms usually start in infancy or early childhood. Patients with the X-linked form of CGD (60-70% of patients) tend to present earlier and have more severe disease than patients with autosomal recessive forms. Most X-CGD develop failure to thrive,recurrentbacteriallymphadenitis and pneumonia due to catalase-positive organism especially staphylococcus, also skin, liver,and other internal organs abscesses, and osteomyelitis. In addition, CGD patients are more subjected to invasive lifethreatening fungal infections that aﬀect the lungs and bones. Another problem with patients diagnosed with CGD is the excessive inﬂammatory reactions leading to granulomatous lesions that typically aﬀects the bladder and gastrointestinal tract.

The primary diagnostic tests used in CGD functionally assess the NADPH complex in stimulated neutrophils.The dihydrorhodamine (DHR) assay is the gold standard for diagnosing CGD.

To the investigator's knowledge this will be the first study in Assiut University Children's Hospital to discuss the clinical characteristics and immunological profile of pediatric patients diagnosed as CGD in Assiut University Children's Hospital. In fact there is defect in data about CGD in upper Egypt .

ELIGIBILITY:
Inclusion Criteria:

Age at enrollment less than18 years. Both genders. Diagnosed as probable CGD.

Exclusion Criteria:

Children above 18 years old. Children not fullfilling the criteria of CGD

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with diagnosed with CGD below 18 yrs
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Immunological Profile and Clinical Characteristics of Children Diagnosed With Chronic Granulomatous Disease | 1 year
  To describe the clinical characteristics and pattern of presentation of patients diagnosed as CGD in Assiut, and to find the most common presenting symptoms.and mention the immunological profile of patients diagnosed with CGD

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] El-Mokhtar MA, Salama EH, Fahmy EM, Mohamed ME. "Clinical Aspects of Chronic Granulomatous Disease in Upper Egypt". Immunol Invest. 2021 Feb;50(2-3):139-151. doi: 10.1080/08820139.2020.1713144. Epub 2020 Jan 22. PMID 31965875
- [Result] Ko SH, Rhim JW, Shin KS, Hahn YS, Lee SY, Kim JG. Genetic analysis of CYBB gene in 26 korean families with X-linked chronic granulomatous disease. Immunol Invest. 2014;43(6):585-94. doi: 10.3109/08820139.2013.825270. PMID 24999735
- [Result] Monies D, Abouelhoda M, AlSayed M, Alhassnan Z, Alotaibi M, Kayyali H, Al-Owain M, Shah A, Rahbeeni Z, Al-Muhaizea MA, Alzaidan HI, Cupler E, Bohlega S, Faqeih E, Faden M, Alyounes B, Jaroudi D, Goljan E, Elbardisy H, Akilan A, Albar R, Aldhalaan H, Gulab S, Chedrawi A, Al Saud BK, Kurdi W, Makhseed N, Alqasim T, El Khashab HY, Al-Mousa H, Alhashem A, Kanaan I, Algoufi T, Alsaleem K, Basha TA, Al-Murshedi F, Khan S, Al-Kindy A, Alnemer M, Al-Hajjar S, Alyamani S, Aldhekri H, Al-Mehaidib A, Arnaout R, Dabbagh O, Shagrani M, Broering D, Tulbah M, Alqassmi A, Almugbel M, AlQuaiz M, Alsaman A, Al-Thihli K, Sulaiman RA, Al-Dekhail W, Alsaegh A, Bashiri FA, Qari A, Alhomadi S, Alkuraya H, Alsebayel M, Hamad MH, Szonyi L, Abaalkhail F, Al-Mayouf SM, Almojalli H, Alqadi KS, Elsiesy H, Shuaib TM, Seidahmed MZ, Abosoudah I, Akleh H, AlGhonaium A, Alkharfy TM, Al Mutairi F, Eyaid W, Alshanbary A, Sheikh FR, Alsohaibani FI, Alsonbul A, Al Tala S, Balkhy S, Bassiouni R, Alenizi AS, Hussein MH, Hassan S, Khalil M, Tabarki B, Alshahwan S, Oshi A, Sabr Y, Alsaadoun S, Salih MA, Mohamed S, Sultana H, Tamim A, El-Haj M, Alshahrani S, Bubshait DK, Alfadhel M, Faquih T, El-Kalioby M, Subhani S, Shah Z, Moghrabi N, Meyer BF, Alkuraya FS. The landscape of genetic diseases in Saudi Arabia based on the first 1000 diagnostic panels and exomes. Hum Genet. 2017 Aug;136(8):921-939. doi: 10.1007/s00439-017-1821-8. Epub 2017 Jun 9. PMID 28600779
- [Result] Boonyawat B, Suksawat Y, Pacharn P, Suwanpakdee P, Traivaree C. X-Linked Chronic Granulomatous Disease: Initial Presentation with Intracranial Hemorrhage from Vitamin K Deficiency in Infant. Case Rep Pediatr. 2018 Jun 24;2018:7041204. doi: 10.1155/2018/7041204. eCollection 2018. PMID 30034904
- [Result] Wakabayashi Y, Jubishi D, Okamoto K, Ikeda M, Tatsuno K, Mizoguchi M, Sato T, Okugawa S, Moriya K. A rare case of a prostatic abscess, bacteremia and chronic granulomatous disease associated with Klebsiella pneumoniae. J Infect Chemother. 2019 May;25(5):365-367. doi: 10.1016/j.jiac.2018.11.015. Epub 2019 Jan 11. PMID 30642769
- [Result] Falcone EL, Holland SM. Invasive fungal infection in chronic granulomatous disease: insights into pathogenesis and management. Curr Opin Infect Dis. 2012 Dec;25(6):658-69. doi: 10.1097/QCO.0b013e328358b0a4. PMID 22964947
- [Result] El Hawary R, Meshaal S, Deswarte C, Galal N, Abdelkawy M, Alkady R, Elaziz DA, Freiberger T, Ravcukova B, Litzman J, Bustamante J, Boutros J, Gaafar T, Elmarsafy A. Role of Flow Cytometry in the Diagnosis of Chronic Granulomatous Disease: the Egyptian Experience. J Clin Immunol. 2016 Aug;36(6):610-8. doi: 10.1007/s10875-016-0297-y. Epub 2016 May 24. PMID 27222152
- [Result] Roesler J, Hecht M, Freihorst J, Lohmann-Matthes ML, Emmendorffer A. Diagnosis of chronic granulomatous disease and of its mode of inheritance by dihydrorhodamine 123 and flow microcytofluorometry. Eur J Pediatr. 1991 Jan;150(3):161-5. doi: 10.1007/BF01963557. PMID 2044584